CLINICAL TRIAL: NCT04673435
Title: Biosynthetic Skin Substitute Versus Frozen Human Cadaver Allograft for Temporary Coverage of Excised Full-thickness Burn Wounds
Brief Title: Permeaderm Versus Homograft for Full-thickness Burns
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol was withdrawn and closed by IRB in April, 2018 prior to enrollment of first patient
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0344
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Full Thickness Burn
Keywords: PermeaDerm; Cadaver skin; full thickness burn; temporary coverage

STUDY DESIGN:
Intervention Model Description: Randomized matched design with application of both study dressings symmetrical or adjacent body sites at the same time.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors (healing time and scar assessments) are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Permeaderm as temporary coverage (Experimental): A: temporary coverage with PermeaDerm until autografting: After randomization of study site, study dressing will be applied as temporary coverage on freshly excised full-thickness burn wounds.
  Interventions: Device: PermeaDerm for temporary coverage
- FHCA as temporary coverage (Active Comparator): B: temporary coverage with FHCA until autografting: After randomization of study site, study dressing will be applied as temporary coverage on freshly excised full-thickness burn wounds.
  Interventions: Device: FHCA for temporary coverage
- Permeaderm over widely meshed autograft (Experimental): C: temporary coverage of widely meshed autograft with PermeaDerm until healing occurs and PermeaDerm can remove
  Interventions: Device: PermeaDerm over autograft
- FHCA over widely meshed autograft (Active Comparator): D: temporary coverage of widely meshed autograft with FHCA until healing occurs
  Interventions: Device: FHCA over autograft

INTERVENTIONS:
Device: PermeaDerm for temporary coverage — See above
  Arms: Permeaderm as temporary coverage
Device: FHCA for temporary coverage — See above
  Arms: FHCA as temporary coverage
Device: PermeaDerm over autograft — See above
  Arms: Permeaderm over widely meshed autograft
Device: FHCA over autograft — see above
  Arms: FHCA over widely meshed autograft

SUMMARY:
Frozen Human Cadaver Allograft (FHCA) is, nowadays, the gold standard for temporary coverage of excised full-thickness burns, but is also very expensive and requires additional personnel and major storage spaces in comparison to other products. The purpose of this study is to determine the extent to which PermeaDerm® dressing promotes wound bed maturation when used as a temporary dressing for excised full-thickness burn wounds. Efficacy and safety in promoting wound bed maturation for successive autografting will be determined through direct comparison to FHCA.

DETAILED DESCRIPTION:
In this prospective, randomized, matched design pilot study, we aim to compare the current standard of care FHCA to PermeaDerm®.

30 patients for each study arm (n total = 60) meeting the inclusion criteria will be enrolled to randomly receive FHCA and PermeaDerm® on two adjacent or symmetric body areas.

Prior to randomization of study areas and application of study dressings, baseline assessments of wound size and burn depth will be performed by the experienced physician and documented using photography and when indicated laser Doppler (Moor Laser Speckle®, Moor Instruments, Devon, UK) measurements. Percentage of graft take and wound healing after removal of the temporary wound dressings and secondary autografting (study arm 1) or after excision and direct autografting with wiedely-meshed autograft and temporary wound dressings as overlay (study arm 2) will be assessed.

Secondary outcomes will include complications such as infections, signs of rejection/non-adherence, fluid accumulation/hematoma beneath dressings and mid- and long-term clinical scar maturation, as assessed by the POSAS and objectively with the DermaLab Combo® device (Cortex Technology ApS, Hadsund, Denmark).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 2 % total body surface area (TBSA) full thickness burned.
* Patients with two adjacent or body symmetrical full thickness burned areas (each ≥ 1 TBSA) and comparable in size (TBSA ± 0.5), that require debridement and autografting.

Exclusion Criteria:

* Time from injury to admission >= 5 days
* Sepsis on admission or clinically suspected infection (as per attending physician)
* Pregnancy or childbearing
* Positive HIV or hepatitis screens
* History of active malignancy
* Patients who do not require surgical debridement and autografting
* Patient with burn injuries originating from other causes (chemical, and frostbite)

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-31 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to heal | up to 8 weeks after initial grafting
  Time until study areas are 95% healed, as rated by blinded assessors based on photographs

SECONDARY OUTCOMES:
Incidence of adherence problems (Arm 2) | up to 21 days after initial surgery
  % of non-adherence at first dressing change
Incidence of adherence problems (Arm 1) | up to 21 days after initial surgery
  % of non-adherence at first dressing change and at time of dressing removal before grafting
Incidence of infections | up to 8 weeks after initial grafting
  Incidence of infection, defined as >10x5 bacteria/g tissue, Only taken when infection suspected.
Rate of fluid/hematoma accumulation | up to 21 days after initial surgery
  % of fluid accumulation/hematoma formation at first dressing change
Cost effectiveness | Until grafting of study sites, within 21 days
  Price per cm square of each study dressing
Scar assessment with Patient and Observer Assessment Scale (POSAS) | Assessed within 4 weeks after 95% wound healing
  Using Patient and Observer Scar Assessment Scale POSAS, what is a composite score that is rating the overall appearance of the scar, based on each single score for rating vascularity, pigmentation, thickness, relief, pliability, surface. Every subscore ranges from 1-10. The composite score is calculated as an average of the subscores. Higher numbers mean worse scarring.
Scar assessment with Patient and Observer Assessment Scale (POSAS) | Assessed between 3 and 9 months after initial admission
  Using Patient and Observer Scar Assessment Scale POSAS, what is a composite score that is rating the overall appearance of the scar, based on each single score for rating vascularity, pigmentation, thickness, relief, pliability, surface. Every subscore ranges from 1-10. The composite score is calculated as an average of the subscores. Higher numbers mean worse scarring.
Scar assessment with Patient and Observer Assessment Scale (POSAS) | Assessed between 9-15 months after initial admission
  Using Patient and Observer Scar Assessment Scale POSAS, what is a composite score that is rating the overall appearance of the scar, based on each single score for rating vascularity, pigmentation, thickness, relief, pliability, surface. Every subscore ranges from 1-10. The composite score is calculated as an average of the subscores. Higher numbers mean worse scarring.
Scarring with DermaLab Combo device: Viscoelasticity | Assessed within 4 weeks after 95% wound healing
  Measured through negative suction and retraction time.
Scarring with DermaLab Combo device: Viscoelasticity | Assessed between 3 and 9 months after initial admission
  Measured through negative suction and retraction time.
Scarring with DermaLab Combo device: Viscoelasticity | Assessed between 9-15 months after initial admission
  Measured through negative suction and retraction time.
Scarring with DermaLab Combo device: Hydration | Assessed within 4 weeks after 95% wound healing
  Measured based on skin conductance.
Scarring with DermaLab Combo device: Hydration | Assessed between 3 and 9 months after initial admission
  Measured based on skin conductance.
Scarring with DermaLab Combo device: Hydration | Assessed between 9-15 months after initial admission
  Measured based on skin conductance.
Scarring with DermaLab Combo device: Pigmentation | Assessed within 4 weeks after 95% wound healing
  Measured based on light absorption of melanin and erythema
Scarring with DermaLab Combo device: Pigmentation | Assessed between 3 and 9 months after initial admission
  Measured based on light absorption of melanin and erythema
Scarring with DermaLab Combo device: Pigmentation | Assessed between 9-15 months after initial admission
  Measured based on light absorption of melanin and erythema
Scarring with DermaLab Combo device: Trans epithermal water loss | Assessed within 4 weeks after 95% wound healing
  Measuring evaporation in g/meter square/hour
Scarring with DermaLab Combo device: Trans epithermal water loss | Assessed between 3 and 9 months after initial admission
  Measuring evaporation in g/meter square/hour
Scarring with DermaLab Combo device: Trans epithermal water loss | Assessed between 9-15 months after initial admission
  Measuring evaporation in g/meter square/hour

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- University of texas Medical Branch Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
data won't be shared